CLINICAL TRIAL: NCT01176721
Title: Transcutaneous Non-invasive Vagus Nerve Stimulation (t-VNS) in the Treatment of Schizophrenia: a Randomized, Controlled, Double Blind, Two-armed Clinical Trial
Brief Title: Transcutaneous Non-invasive Vagus Nerve Stimulation (t-VNS) in the Treatment of Schizophrenia
Acronym: 02VNS2009
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: cerbomed GmbH (Industry)
Collaborators: Institut fuer anwendungsorientierte Forschung und klinische Studien GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 02VNS2009
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Schizophrenia
Keywords: schizophrenic disorders; psychosis; psychotic; dementia; delusional; delusions; hallucinations; residual-type schizophrenia; illusions; split mind; mental health disorder; schizoid; paranoid-type schizophrenia; disorganized-type schizophrenia; undifferentiated-type schizophrenia; catatonic-type schizophrenia; mental illness; tardive dyskinesia; neuroleptic malignant syndrome; NMS; antipsychotics; atypical antipsychotics; psychosocial treatments; rehabilitation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mental Disorders; Dementia; Delusions; Hallucinations; Illusions; Schizophrenia, Paranoid; Schizophrenia, Disorganized; Schizophrenia, Catatonic; Tardive Dyskinesia; Neuroleptic Malignant Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- t-VNS verum (Active Comparator): Active stimulation of the left auricle by t-VNS
  Interventions: Device: t-VNS verum
- Sham (Placebo Comparator): Sham-simulation of the left auricle by the t-VNS device.
  Interventions: Device: t-VNS placebo

INTERVENTIONS:
Device: t-VNS verum — Active stimulation of the left auricle by t-VNS
  Arms: t-VNS verum
Device: t-VNS placebo — Sham stimulation of the left auricle with the t-VNS device
  Arms: Sham

SUMMARY:
Randomized, controlled, double-blind, two-armed clinical investigation to show the efficacy and safety of transcutaneous vagus nerve stimulation (t-VNS), applied at the left auricle, in schizophrenia.

Study hypothesis: t-VNS may improve negative symptoms, depressive symptoms, cognitive impairment,and aggressive behavior of treated schizophrenia patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a schizophrenic disorder (F20 according to ICD-10),duration of disease ≥ 12 months
* Appliance of the t-VNS® medical device according to the manual

Exclusion Criteria:

* Improvent of the PANSS score within the period of 2 - 4 weeks from screening to the baseline
* Pregnancy
* Bronchial asthhma in medical history
* clinically relevant internistic, neurological or psychiatric diseases
* abuse of drugs or alcohol until 4 weeks to enrollment
* Traumatic brain injury in medical history as well as invasive and non-invasive methods of treatment (e.g. tumor surgery (Gammma knife surgery))
* indication of structural impairment of the basal ganglia or the brain stem
* malformations of the pinna
* further circumstances that at the discretion of the investigator will not allow to include the subject into the clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2011-07 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy of t-VNS in schizophrenia | 24 weeks

SECONDARY OUTCOMES:
Recording of clinical performance of t-VNS in schizophrenia | 24 weeks
  self rating:
  * BDI
  * Fagerström
  rating by investigator
  * UKU
  * SANS
  * CDSS
  * MARDS
  * HAMD-21
  * CGI
  * PSP
  * SWN_K
  * St. Hans
  * VLMT
  * TMT-B
  * TMT-A
  * RWT
  * Corsi Block Tapping
  * Zahlennachsprechen
  * MWT-B
  * EKT
  * HR
  * dTMS

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Department of Psychiatry and Psychotherapy, Ludwig-Maximilians-Universitaet Muenchen, Munich, Bavaria
  - Departement of Psychiatry and Psychotherapy, University Hospital of Goettingen, Göttingen, Lower Saxony